CLINICAL TRIAL: NCT02782780
Title: Pilot Test of Telephone-Delivered Cognitive Behavioral Therapy for Insomnia for Veterans With Gulf War Illness
Brief Title: Cognitive Behavioral Therapy for Insomnia for Gulf War Illness
Acronym: CBTi GWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPLD-12-15F; I21CX001428 (NIH)
Record Dates: First submitted 2016-05-23; First posted 2016-05-25 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Gulf War Illness; Insomnia
Keywords: insomnia; insomnia disorder; Gulf War Illness; Chronic Multisymptom Illness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBTi (Experimental): CBTi is a multicomponent treatment that seeks to teach patients about sleep and the factors that affect sleep as well as to work with the patient toward altering sleep habits to increase sleep propensity and regularity. Specifically, participants will receive 8 weekly individual sessions of CBTi according to the VA CBTi protocol. The investigators will follow the semi-structured approach to treatment described in the VA CBTi protocol, which allows the case conceptualization to drive the order in which treatment components are introduced.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTi)
- Monitor Only (No Intervention): Study participants who are randomized to the Monitor Only (MO) control group will be followed for 8 weeks of usual care (i.e., they will be advised to continue doing whatever they were doing to manage their GWI and insomnia symptoms without change dosage or frequency of treatment). Participants randomized to the Monitor Only condition will have the option of receiving CBTi delivered by telephone, at no cost to them, upon completion of post-study procedures.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTi) — CBTi is a multicomponent treatment that seeks to teach patients about sleep and the factors that affect sleep (e.g., homeostatic regulation, circadian rhythm, age, social and work schedule) and to work with the patients toward minimizing unwanted arousal at bedtime and altering sleep habits to increase sleep propensity and regularity. The intervention is 8-weeks long.
  Other Names: CBTi
  Arms: CBTi

SUMMARY:
Sleep disturbance is a common complaint of Veterans with Gulf War Illness (GWI). Because there is clinical evidence that sleep quality influences pain, fatigue, mood, cognition, and daily functioning, this study will investigate whether a type of behavioral sleep treatment called Cognitive Behavioral Therapy for Insomnia (CBTi) can help Gulf War Veterans with GWI. CBTi is a multicomponent treatment where patients learn about sleep and factors affecting sleep as well as how to alter habits that may impair or even prevent sleep. The investigators hypothesize that helping Gulf War Veterans learn how to achieve better sleep with CBTi may also help to alleviate their other non-sleep symptoms of GWI.

DETAILED DESCRIPTION:
Insomnia is common among Veterans with Gulf War Illness (GWI). Moreover, untreated insomnia is associated with significant medical and psychiatric morbidity. Cognitive Behavioral Therapy for Insomnia (CBTi) is a multicomponent treatment that seeks not only to teach patients about sleep and factors affecting sleep (e.g., circadian rhythm, age, social and work schedule) but the therapist will also to work with the patient toward minimizing unwanted arousal at bedtime and altering sleep habits to increase sleep propensity and regularity.

Because many Veterans with GWI suffer from a profound loss of physical and functional status that may prevent them from participating in treatments that require regular clinic visits, the proposed study will deliver CBTi by telephone to extend this effective form of behavioral sleep medicine to Veterans who have chronic illnesses and disabilities and/or who live in rural areas with limited access to trained CBTi providers. Recent studies suggest that telephone-delivered CBTi is as effective as CBTi delivered in-person.

The proposed trial will examine the efficacy of telephone-delivered CBTi for alleviating sleep and non-sleep GWI symptoms in a two-arm randomized controlled trial. Veterans who have GWI and persistent insomnia disorder will be randomized to a group that will receive CBTi right away or to a group that will receive treatment-as-usual (i.e., the control group). Veterans randomized to the control group will have the option of receiving telephone-delivered CBTi upon completion of post-treatment assessments. The primary outcomes will be effect sizes base on within-group comparisons of pre-to-post-treatment change and maintenance of treatment effects at 6 months in the CBTi group.

ELIGIBILITY:
Inclusion Criteria:

* Deployed to the Gulf Theater of operations, as defined by 38 CFR 3.317 in the years 1990-1991, in accordance with the inclusion/exclusion criteria set forth in the federal definition of Gulf War Illness as used for the Gulf War Registry.

  * This will be confirmed through VA records or by asking veterans to provide a copy of their DD214.
* Have Gulf War Illness (GWI) according to the Kansas case definition.

  * GWI symptom will be assessed with the Kansas Gulf War Military History and Health Questionnaire.
* Have an Insomnia Severity Index score greater than or equal to 14.

Exclusion Criteria:

* Have conditions or substances that may be associated with comorbid insomnia independent of GWI status, including:

  * a lifetime history of any psychiatric disorder with psychotic features
  * bipolar disorder
  * panic disorder
  * obsessive-compulsive disorder
  * alcohol or substance dependence
  * a history of alcohol or substance abuse within the past year
* Currently exposed to recurrent trauma or have been exposed to a traumatic event within the past 3 months.
* Pregnancy (because insomnia will worsen after 8 weeks).
* Prominent suicidal or homicidal ideation.
* History of sleep restriction therapy or cognitive restructuring therapies of beliefs related to sleep.
* Subjects concurrently enrolled in another clinical trial.
* Veterans who work night shifts or have extreme morning or evening tendencies as described below will be excluded in order to avoid the impact of circadian factors on evaluating insomnia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda L. Chao, PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from October 2016 to July 2019 by flyers, on-line recruitment, direct mailings to past GW Veteran participants and those on a list provided by the Department of Defense Manpower Data Reporting Center.
  Of the 165 participants enrolled/consented, 27 did not undergo/complete the clinical assessment interview, 42 were ineligible after the clinical assessment interview, and 11 did not complete baseline assessment. Therefore, only 85 participants were randomized.
Pre-assignment Details: During the first phase of screening, veterans participated in a brief telephone interview to inquire about inclusion/exclusion criteria and to determine probable GWI/CMI and insomnia diagnoses. Only participants who passed the initial telephone eligibility screening were invited to undergo a second round of clinical screening to assess for mental health disorders and other exclusionary conditions (e.g., untreated sleep apnea and restless legs syndrome).
Period: Overall Study
Arm/Group | Monitor Only | CBTi
Started | 46 | 39
Completed | 39 | 32
Not Completed | 7 | 7
Not completed — dropped out after randomization. | 7 | 5
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monitor Only | CBTi | Total
Number analyzed (Participants) | 46 | 39 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (6) | 55 (7) | 54.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 36 | 28 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 11 | 19
  White | 36 | 25 | 61
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 39 | 85

OUTCOME MEASURES:

1. Primary Outcome: Gulf War Illness Symptom Severity Index
Description: Due to its novelty, complexity, and variability, no single measure of severity addresses all possible presentations of Gulf War Illness (GWI). Therefore, we used the symptom portion of the Kansas Gulf War Military History and Health Questionnaire to query about fatigue/sleep problems, somatic pain, skin abnormalities, gastrointestinal, respiratory, and neurologic/cognitive/mood symptoms, based on the Kansas GWI and CDC CMI case definition. To assess current GWI symptoms, participants will be asked about the absence (0), presence, and severity (1=mild; 2=moderate; 3=severe) of the symptoms over the past 2 weeks instead of over the past 6-months. Score range: 0-87; higher scores = more symptoms and/or more severe symptoms.
Time Frame: At baseline, after 8 weeks of study participation in all subjects, in subjects randomized to CBTi, 6 months after study participation
Population: 32 of 39 participants randomized to CBTi completed treatment; only 28 of these participants completed the 6-month follow-up assessment.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Monitor Only | CBTi
Number analyzed (Participants) | 46 | 39
score on a scale
  Baseline | 67 [53 to 78] | 67 [58 to 82]
  Post-treatment | 61 [50 to 78] | 49 [44 to 62]
  6-month follow-up: number analyzed (Participants) | 0 | 28
  6-month follow-up |  | 54 [49 to 66]
Statistical Analysis 1: Comparison: Monitor Only vs CBTi; Test type: Superiority — Linear mixed models with random effects for subjects were used to analyze all available data for the intent-to-treat analysis. Because sex was used as a stratification variable in the randomization procedure, it was not included as a covariate the analyses; p < 0.01, Mixed Models Analysis — Test of treatment effect: t(91.6)=3.21
Statistical Analysis 2: Comparison: CBTi; Test type: Superiority; p < 0.001, Mixed Models Analysis — Baseline vs. 6-month follow-up in CBTI group: t(92.3)=4.10; Planned contrasts following the mixed models were used to compare baseline data to 6-month follow-up data in the CBTI group

2. Primary Outcome: Insomnia Severity Index (ISI)
Description: The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia in the last month. The dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. Higher scores indicate more severe insomnia. This outcome will be measured at 8 weeks in both the CBTi and monitor-only groups and at 6 months in subjects randomized to CBTi.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Monitor Only | CBTi
Number analyzed (Participants) | 46 | 39
score on a scale
  Baseline | 19.0 [16.0 to 24.0] | 21.0 [18.0 to 24.0]
  post-treatment | 19.0 [13.5 to 22.0] | 10.0 [6.0 to 15.0]
  6-month follow-up: number analyzed (Participants) | 0 | 28
  6-month follow-up |  | 13.0 [7.0 to 18.0]
Statistical Analysis 1: Comparison: Monitor Only vs CBTi; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis — test of treatment effect: t(94.7)=6.10
Statistical Analysis 2: Comparison: CBTi; To compare baseline data to 6-month follow-up data in the CBT-I group, planned contrasts following the mixed models were used; Test type: Superiority; p < 0.001, Mixed Models Analysis — baseline vs. 6-month follow-up in CBTI group: t(94)=6.67; [statistical method as in outcome 1, analysis 2]

3. Secondary Outcome: Fatigue Severity Scale (FSS)
Description: The FSS is a 9-item questionnaire reflecting the consequences of fatigue. It gives a single score (range 0-7, high scores represent high levels of fatigue). A score of 4 has been described as the cutoff for clinical fatigue. This outcome will be measured at baseline, after 8 weeks in both the CBTi and monitor-only groups and at 6 months in subjects randomized to CBTi.
Time Frame: Baseline, after 8 weeks of study participation in all subjects, in subjects randomized to CBTi, 6 months after study participation
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Monitor Only | CBTi
Number analyzed (Participants) | 46 | 39
score on a scale
  Baseline | 5.06 [3.47 to 5.78] | 5.56 [4.67 to 6.28]
  Post-treatment | 5.11 [3.22 to 5.83] | 3.44 [2.89 to 5.03]
  6-month follow-up: number analyzed (Participants) | 0 | 28
  6-month follow-up |  | 3.67 [2.78 to 5.44]
Statistical Analysis 1: Comparison: Monitor Only vs CBTi; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; test of treatment effect: t(104)=3.40
Statistical Analysis 2: Comparison: CBTi; Test type: Superiority; p < 0.001, Mixed Models Analysis — Baseline vs. 6-month follow-up in CBTi group: t(91.6)=4.37; [statistical method as in outcome 1, analysis 2]

4. Secondary Outcome: Brief Pain Inventory (BPI) - Pain Interference
Description: The BPI is a 17-item self-rating scale assessing demographic data, use of medications, as well as sensory, and reactive components of pain. The BPI measures two domains: pain intensity (severity) and the impact of pain on functioning (interference). The score range for BPI-Severity is 0-10, higher score = more severe/intense pain. The range for BPI-interference is 0-10, higher score = greater impact of pain on function.
  This outcome will be measured at baseline, after 8 weeks in both the CBTi and monitor-only groups and at 6 months in subjects randomized to CBTi.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Monitor Only | CBTi
Number analyzed (Participants) | 46 | 39
score on a scale
  Baseline | 4.29 [2.46 to 6.68] | 5.86 [3.79 to 7.29]
  Post-treatment | 4.57 [2.07 to 6.86] | 4.29 [1.57 to 5.57]
  6-month follow-up: number analyzed (Participants) | 0 | 28
  6-month follow-up |  | 4.29 [1.64 to 6.64]
Statistical Analysis 1: Comparison: Monitor Only vs CBTi; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.05, Mixed Models Analysis; test of treatment effect: t(99.9)=2.09
Statistical Analysis 2: Comparison: CBTi; Planned contrasts following the mixed models were used to compare baseline data to 6-month follow-up data in the CBTi group; Test type: Superiority; p < 0.01, Mixed Models Analysis; Baseline vs. 6-month follow-up in CBTi group: t(92.1)=2.56

5. Secondary Outcome: Brief Pain Inventory (BPI) - Pain Severity
Description: as for outcome 4
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Monitor Only | CBTi
Number analyzed (Participants) | 46 | 39
score on a scale
  Baseline | 4.12 [2.88 to 6.75] | 5.00 [3.38 to 6.50]
  Post-treatment | 4.25 [2.88 to 5.75] | 5.25 [3.00 to 5.75]
  6-month follow-up: number analyzed (Participants) | 0 | 28
  6-month follow-up |  | 5.00 [3.00 to 6.00]
Statistical Analysis 1: Comparison: Monitor Only vs CBTi; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.991, Mixed Models Analysis; Test of treatment effect: t(110)=-0.41
Statistical Analysis 2: Comparison: CBTi; Test type: Superiority; p = 0.41, Mixed Models Analysis — Baseline vs. 6-month follow-up in CBTi group: t(91.8)=0.94; [statistical method as in outcome 1, analysis 2]

6. Secondary Outcome: Multiple Abilities Self-Report Questionnaire (MASQ)
Description: The MASQ is a 38-item self-report measure of cognitive function compared to same age peers across 5 domains (i.e., verbal memory, attention, language, visual memory, visuo-perceptual ability). Score range: 38-190. Higher scores = greater cognitive dysfunction.
  This outcome will be measured at baseline, after 8 weeks in both the CBTi and monitor-only groups and at 6 months in subjects randomized to CBTi.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Monitor Only | CBTi
Number analyzed (Participants) | 46 | 39
score on a scale
  Baseline | 64 [39 to 77] | 61 [44 to 76]
  Post-treatment | 68 [42 to 89] | 55 [37 to 69]
  6-month followup: number analyzed (Participants) | 0 | 28
  6-month followup |  | 54 [44 to 77]
Statistical Analysis 1: Comparison: Monitor Only vs CBTi; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.05, Mixed Models Analysis; Test of treatment effect: t(83.7)=2.51
Statistical Analysis 2: Comparison: CBTi; Test type: Superiority; p = 0.49, Mixed Models Analysis — Planned contrasts following the mixed models were used to compare baseline data to 6-month follow-up data in the CBTi group; Baseline vs. 6-month follow-up in CBTi group: t(90.9)=0.27

7. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS), Anxiety
Description: The HADS will be used to assess anxiety and depressive symptoms. The HADS is widely used in community settings and in primary care and not just in "hospitals." The range for HADS-anxiety measure is 0-21. Higher scores = more anxiety.
  This outcome will be measured at baseline, after 8 weeks in both the CBTi and monitor-only groups and at 6 months in subjects randomized to CBTi.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Monitor Only | CBTi
Number analyzed (Participants) | 46 | 39
score on a scale
  Baseline | 10.5 [6.2 to 13.8] | 12.5 [9.2 to 14.0]
  Post-treatment | 11.0 [7.0 to 15.5] | 8.0 [5.0 to 11.0]
  6-month follow-up: number analyzed (Participants) | 0 | 28
  6-month follow-up |  | 9.0 [6.5 to 11.0]
Statistical Analysis 1: Comparison: Monitor Only vs CBTi; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.01, Mixed Models Analysis; test of treatment effect: t(105)=4.55
Statistical Analysis 2: Comparison: CBTi; Test type: Superiority; p < 0.01, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; Baseline vs. 6-month follow-up in CBTi group: t(91.3)=3.23

8. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS), Depression
Description: The HADS will be used to assess anxiety and depressive symptoms. The HADS is widely used in community settings and in primary care and not just in "hospitals." The range for HADS-depression measure is 0-21. Higher scores = more anxiety.
  This outcome will be measured at baseline, after 8 weeks in both the CBTi and monitor-only groups and at 6 months in subjects randomized to CBTi.
Time Frame: as for outcome 3
Population: Only 28 participants completed the 6-month assessments.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Monitor Only | CBTi
Number analyzed (Participants) | 46 | 39
score on a scale
  Baseline | 9.0 [5.2 to 11.8] | 9.5 [7.0 to 12.0]
  Post-treatment | 9.0 [5.5 to 11.0] | 4.0 [2.0 to 8.0]
  6-month follow-up: number analyzed (Participants) | 0 | 28
  6-month follow-up |  | 6.0 [3.0 to 9.0]
Statistical Analysis 1: Comparison: Monitor Only vs CBTi; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Test of treatment effect: t(91.6)=3.37
Statistical Analysis 2: Comparison: CBTi; Test type: Superiority; p < 0.001, Mixed Models Analysis — Baseline vs. 6-month follow-up in CBTi group: (92.1)=3.64; [statistical method as in outcome 1, analysis 2]

9. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI is a self-report measure that provides a subjective assessment of sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sedative-hypnotics, and daytime energy. This index is widely used and has been validated by polysomnography. The score range for the PSQI is 0 to 21, with the higher scores indicating worse sleep quality.This outcome will be measured at baseline, after 8 weeks in both the CBTi and monitor-only groups and at 6 months in subjects randomized to CBTi.
Time Frame: as for outcome 3
Population: Only 28 of the participants randomized to CBTi completed the 6-month follow-up assessment.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Monitor Only | CBTi
Number analyzed (Participants) | 46 | 39
score on a scale
  Baseline | 12.0 [9.2 to 14.8] | 11.0 [9.0 to 15.0]
  Post-treatment | 11.0 [8.5 to 13.0] | 8.0 [3.0 to 9.0]
  6-month follow-up: number analyzed (Participants) | 0 | 28
  6-month follow-up |  | 7.0 [5.0 to 10.5]
Statistical Analysis 1: Comparison: Monitor Only vs CBTi; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Test of treatment effect: t(99.2)=5.45
Statistical Analysis 2: Comparison: CBTi; Test type: Superiority; p < 0.001, Mixed Models Analysis — Baseline vs. 6-month follow-up in CBTi group: t(93.4)=6.06; [statistical method as in outcome 1, analysis 2]

10. Secondary Outcome: Sleep Efficiency (SE)
Description: Sleep Efficiency, as determined by self-reported sleep diary, is the total sleep time (TST) divided by the time in bed, multiplied by 100. Good sleepers have high sleep efficiency because they are asleep the majority of time they spend in bed. Insomniacs tend to have low sleep efficiency because they spend a lot of time awake while they are in bed (tossing and turning).
  This outcome will be measured at baseline, after 8 weeks in both the CBTi and monitor-only groups and at 6 months in subjects randomized to CBTi.
Time Frame: as for outcome 3
Population: Only 28 of the participants randomized to CBTi completed the 6-month assessment.
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Monitor Only | CBTi
Number analyzed (Participants) | 46 | 39
percent
  Baseline | 82 [74 to 89] | 83 [74 to 88]
  Post-treatment | 78 [73 to 89] | 94 [90 to 95]
  6-month follow-up: number analyzed (Participants) | 0 | 28
  6-month follow-up |  | 91 [89 to 94]
Statistical Analysis 1: Comparison: Monitor Only vs CBTi; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; test of treatment effect: t(76.9)=-4.20
Statistical Analysis 2: Comparison: CBTi; Test type: Superiority; p < 0.001, Mixed Models Analysis — Baseline vs. 6-month follow-up in CBTi group: t(33.1)=6.52; [statistical method as in outcome 1, analysis 2]

11. Secondary Outcome: Minutes of Wake After Sleep Onset (WASO)
Description: Wake After Sleep Onset is the amount of time that a person is awake time during the night, as recorded in a self-report sleep diary. Insomniacs tend to have greater WASO than good sleepers because they wake up a lot in the middle of the might.
  This outcome will be measured at baseline, post-treatment in both the CBTi and monitor-only groups and at 6 months in subjects randomized to CBTi.
Time Frame: Baseline and after 8 weeks of study participation in all subjects; in subjects randomized to CBTi, 6 months after study participation
Population: Only 28 of the participants randomized to CBTi completed the 6-month follow-up assessment.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Monitor Only | CBTi
Number analyzed (Participants) | 46 | 39
minutes
  Baseline | 25 [11 to 43] | 31 [19 to 53]
  Post-treatment | 33 [18 to 57] | 7 [4 to 22]
  6-month follow-up: number analyzed (Participants) | 0 | 28
  6-month follow-up |  | 20 [11 to 27]
Statistical Analysis 1: Comparison: Monitor Only vs CBTi; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Test of treatment effect: t(75.6)=4.33
Statistical Analysis 2: Comparison: CBTi; Test type: Superiority; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; Baseline vs. 6-month follow-up in CBTi group: t(34.4)=4.75

12. Secondary Outcome: Sleep Latency (SL)
Description: Sleep latency (SL) is the amount of time that it takes someone to fall asleep. Participants will be asked to estimate this time in their sleep diaries. Good sleepers tend to have low sleep latencies because they can fall asleep quickly. Insomniacs tend to have longer sleep latencies because it takes them a long time to fall asleep.
  This outcome will be measured at baseline, after 8 weeks in both the CBTi and monitor-only groups and at 6 months in subjects randomized to CBTi.
Time Frame: as for outcome 3
Population: Only 28 participants randomized to CBTi completed the 6-month follow-up.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Monitor Only | CBTi
Number analyzed (Participants) | 46 | 39
minutes
  Baseline | 22 [15 to 44] | 22 [13 to 34]
  Post-treatment | 24 [14 to 46] | 10 [7 to 12]
  6-month follow-up: number analyzed (Participants) | 0 | 28
  6-month follow-up |  | 12 [7 to 16]
Statistical Analysis 1: Comparison: Monitor Only vs CBTi; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; Test of treatment effect: t(75.1)=3.91
Statistical Analysis 2: Comparison: CBTi; Test type: Superiority; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; Baseline vs. 6-month in CBTi group: t(34.5)=4.39

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Monitor Only | CBTi
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/39
Other Adverse Events (participants affected / at risk) | 0/46 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT02782780/Prot_SAP_ICF_000.pdf